CLINICAL TRIAL: NCT06842290
Title: Effect of Botulinum Toxin -A Injection in Mentalis Muscle with Coronally Advanced Flap and De-epithelized Free Gingival Graft in Treatment of RT1 , RT2 Gingival Recession _Randomized Control Trial
Brief Title: Effect of Botulinum Toxin a Injection in Treatment of Recession RT1 and RT2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mayar Mostafa Tawfik Ali, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER3,3,2
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): In this arm principal investigator will preform coronally advanced flap with De-epithelized free gingival graft then will inject Botulinum toxin-A in Mentalis muscle after suturing
  Interventions: Procedure: Botulinum toxin-A injection
- Control arm (Active Comparator): In this arm no injection will be applied only coronally advanced flap with De-epithelized free gingival graft alone
  Interventions: Procedure: Coronally advanced flap

INTERVENTIONS:
Procedure: Botulinum toxin-A injection — Botulinum toxin-A Injection Mentalis muscle in lower anterior teeth
  Arms: Intervention arm
Procedure: Coronally advanced flap — Coronally Advanced Flap andDe-epithelized Free Gingival Graft
  Arms: Control arm

SUMMARY:
The goal of this study type: clinical trial] is to learn the effect of Botulinum Toxin _A injection in treatment of RT1andRT2 Gingival recession in lower anterior teeth .

Primary outcome is keratinzed tissue width. Researchers will compare Coronally Advanced flap with De-epithelized free gingival graft and Botulinum toxin-A injection in Mentalis muscle with coronally advanced flap with De-epithelized free gingival graft alone .

The outcome will be measured at baseline, after 3 months and after 6 mobths _medical history

* 3 mm horizontal incisions, then two vertical incisions
* deepitheliztion of anatomical papillae
* superficial and deep incisions
* harvesting DFGG
* Suturing
* BOTOX injection

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple RT1, RT2 GR patient
* patients ≥18 years
* systemically healthy, full mouth plaque score, full mouth bleeding score ≤ 15% after phase I therapy
* clinical indication and/or patient request for recession coverage
* well motivated patients, maintaining oral hygiene throughout study

Exclusion Criteria:

* Pregnant or lactating women
* Smokers' patients
* Teeth with cervical restorations/abrasion.
* Patients had a systemic condition affect blood components and healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-04 (Estimated); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Keratinized tissue width | Measured at baseline ,3months ,6 months